CLINICAL TRIAL: NCT02588391
Title: Randomized Controlled Trial of Executive Function Training in Preterm Children at Risk for Inattention, Hyperactivity and Executive Function Impairment
Brief Title: Brain Training in Preterm Children at Risk for Inattention, Hyperactivity, and Executive Function Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Irene M. Loe, MD, Principal Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 30874; K23HD071971 (NIH)
Record Dates: First submitted 2015-10-26; First posted 2015-10-27 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Premature Birth
Keywords: premature birth; executive function; preschool
MeSH Terms: conditions — Premature Birth | interventions — Cognitive Training; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active Brain Training (Experimental): The children in this arm receive one type of "Brain Training" with online computer games that actively matches their skill level.
  Interventions: Behavioral: Brain Training (Active)
- Passive Brain Training (Experimental): The children in this arm receive one type of "Brain Training" with online computer games that are at a consistent skill level.
  Interventions: Behavioral: Brain Training (Passive)
- Cross-over (Other): Following completion of the 6-month follow-up sessions after completion of "Brain Training", each group is allowed to cross-over to the other arm of "Brain Training" (open-label extension).
  Interventions: Behavioral: Brain Training (Active or Passive)

INTERVENTIONS:
Behavioral: Brain Training (Active) — Online computer games targeting attention, EF, and problem-solving match the child's skill level.
  Arms: Active Brain Training
Behavioral: Brain Training (Passive) — Online computer games targeting attention, EF, and problem solving are set to a consistent level.
  Arms: Passive Brain Training
Behavioral: Brain Training (Active or Passive) — Online computer games targeting attention, EF, and problem-solving either match the child's level or are set to a consistent level depending on which version the child has already completed.
  Arms: Cross-over

SUMMARY:
The purpose of this study is to determine if different forms of child-friendly, computer-based puzzles and games ("brain training") targeting executive function (EF) skills (i.e., thinking, problem-solving) result in improvements in EF in preschool children at risk for EF problems due to premature birth. The investigators hypothesize that children receiving active "brain training" will show greater improvements in EF and related skills immediately after treatment than children receiving passive "brain training." The investigators are also interested in whether any improvements in EF and related skills occur or are maintained at 3 and 6 months after completion of brain training.

DETAILED DESCRIPTION:
Detailed description:

* Investigators will talk to you by telephone to determine if your child might be eligible for the study.
* Children complete two baseline testing sessions to evaluate executive function (EF) and related skills
* Parents complete a packet of information, including questionnaires about the child's behavior, EF, and functional skills.
* After completion of the baseline testing, we will inform you of eligibility for the "Brain Training" phase.
* During "Brain Training" children play online computer games for 25-30 minutes/day (can range from 15-45 minutes/day depending on your child's attention, training version received, number and length of breaks needed), 5 days a week, for 5-7 weeks to complete a total of 25 sessions.
* Children return for 3 more time points, immediately after the completion of "Brain Training" (1 session), and also at 3 months (1 session) and 6 months (2 sessions) after completion of "Brain Training."

ELIGIBILITY:
Inclusion Criteria:

* Age 4 or 5 years
* Born prematurely at <33 weeks gestation
* Able to comprehend task instructions
* EF impairment on standardized questionnaire (t-score of 60 or greater) or EF battery (lower quartile)

Exclusion Criteria:

* Major neurosensory impairment (i.e., blind, deaf) or technology dependence (i.e., ventilator dependent) that interferes with testing
* Genetic syndrome
* Inability to comprehend task instructions

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2015-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline on Executive Function Composite Measure at 2 months | 2 months
  EF composite measured post "Brain Training."

SECONDARY OUTCOMES:
Change from baseline on Executive Function Composite Measure at 5 months | 5 months
  EF composite measured 3-months post "Brain Training" and 5 months from baseline
Change from baseline on Executive Function Composite Measure at 8 months | 8 months
  EF composite measured 6-months post "Brain Training" and 8 months from baseline
Change from baseline on Early Academic Skills Measures at 8 months | 8 months
  Composite scores from standardized measures of pre-academic skills and early literacy and numeracy measures at 6-months post "Brain Training" and 8 months from baseline
Change from 8-month Executive Function Composite Measure at 10 months (cross over groups) | 2 months
  Children who cross-over to the other "Brain Training" intervention arm after the 8 month follow-up visit, will be re-assessed at the completion of the alternate version of "Brain Training"

CONTACTS AND LOCATIONS:
Overall Officials: Irene M Loe, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States